CLINICAL TRIAL: NCT02908347
Title: A Randomized (1:1), Double-blind, Parallel, Placebo-controlled Exploratory Pilot Study to Evaluate the Safety, Pharmacokinetics and Efficacy of Systemic (po) Application of MP1032 in Patients With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Study to Evaluate Safety and Efficacy of Oral MP1032 in Psoriasis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MetrioPharm AG (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP1032-CT02
Record Dates: First submitted 2016-06-23; First posted 2016-09-20 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Psoriasis; Plaque Psoriasis
Keywords: Plaque psoriasis; chronic; moderate; severe; Plaque
MeSH Terms: conditions — Psoriasis; Bronchiolitis Obliterans Syndrome; Lymphoma, Follicular; Plaque, Amyloid | interventions — sodium luminolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MP1032 (Experimental): Test Product:
  100 mg MP1032 (= 2 capsules a 50 mg) are provided orally twice daily for 42 days
  Interventions: Drug: MP1032
- Placebo (Experimental): Placebo to MP1032:
  2 capsules of Placebo are provided orally twice daily for 42 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MP1032 — hard gelatine capsules containing 50 mg MP1032 as active ingredient
  Arms: MP1032
Drug: Placebo — hard gelatine capsules without active ingredient
  Arms: Placebo

SUMMARY:
This Phase IIa study is designed to assess the safety, tolerability and pharmacokinetics of oral MP1032 in patients with moderate to severe psoriasis over a period of 6 weeks. Secondary endpoints to evaluate clinical parameters for psoriasis during the 6 week treatment period and a 4-week follow up will provide an opportunity to perform a first assessment of oral MP1032's clinical efficacy in the treatment of moderate to severe psoriasis.

The study population will consist of 44 enrolled (40 completed) patients with moderate to severe chronic plaque psoriasis. Patients must be able to provide written consent and meet all the inclusion criteria and none of the exclusion criteria.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, parallel, placebo-controlled exploratory pilot study to evaluate safety, pharmacokinetics and efficacy of systemic oral (po) administration of 100 mg MP1032 bid in adult patients with moderate to severe chronic plaque psoriasis.

The study design consists of a 28-day screening/run-in period, a 42-day treatment period, 1 day for the End of Treatment visit, and a 28-day follow-up period. Forty-four patients who meet the entry criteria will be randomized on Day 1 in a 1:1 ratio to receive either 100 mg MP1032 or placebo orally twice daily for 42 days. The goal is to have 40 patients (20 in each treatment group) complete the study.

Pharmacokinetic sampling will occur on 3 designated study days. Safety will be monitored from the signing of the informed consent form (ICF) until the last follow-up visit on Day 71.

Efficacy will be assessed on 6 designated study days using the following assessments: PASI, PGA, DLQI, mNAPSI, and EQ-5D 5L (VAS).

ELIGIBILITY:
Inclusion Criteria:

1. Participants legally competent to sign and give informed consent.
2. Adult male and female patients aged 18 to 65 years with chronic plaque psoriasis:

   1. PASI score > 10 at screening and
   2. Disease duration of ≥ 6 months at the initiation of study medication.
3. Body Mass Index (BMI) between 18.5 and 34.9 kg/m2.
4. Diagnosis of chronic plaque psoriasis confirmed by a dermatologist/physician.
5. Women of childbearing potential (WCBP) must have a negative urine pregnancy test at Screening (Visit 1). In addition, sexually active WCBP must agree to use 2 forms of adequate contraception throughout the trial.
6. Post-menopausal women with spontaneous amenorrhea for at least 12 months and serum levels follicle stimulating hormone (FSH) Levels indicating post-menopausal state as per local laboratory reference ranges. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2 to 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study. Sterilized women may be included.
7. Patients must meet the following clinical laboratory criteria:

   1. White blood cell count ≥ 3.5 x 10^9/L
   2. Platelet count ≥ 100 x 10^9/L
   3. Serum creatinine ≤ 1.5 x upper limit of normal (ULN); estimated glomerular filtration rate > 60 mL/min
   4. Total bilirubin ≤ 1.5 x ULN
   5. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 1.5 x ULN
   6. Hemoglobin ≥ lower limit of normal as per local laboratory reference ranges for women and men accordingly
   7. No coagulopathy (International Normalized Ratio [INR] < 1.5).
8. Patients agree not to increase normal sun exposure during the course of the study.
9. Patients are able to swallow 2 small capsules during each administration.
10. Patients are considered reliable and capable of adhering to the protocol (eg, able to understand and complete diaries), visit schedule, or medication intake according to the judgment of the Investigator.

Exclusion Criteria:

1. Patients with non-plaque form of psoriasis (erythrodermic, guttate, pustular or palmo plantar psoriasis; severe form of psoriasis arthritis, inverse form of psoriasis). Mild to moderate cases of psoriasis arthritis are allowed provided there is no impact on study objectives as determined by the Investigator.
2. Patients with drug-induced psoriasis.
3. Evidence of skin conditions at the time of screening visit other than psoriasis that would interfere with evaluations of the effect of study medication on psoriasis.
4. Patients with any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing the informed consent form.
5. Pregnant or lactating females or females planning to become pregnant during the study and/or within 28 days following the last dose of study medication.
6. Male patients planning a partner pregnancy or sperm donation during the study or within 3 months following the last dose of study medication.
7. Known allergies to mannitol, macrophage modulators, and gelatin.
8. Patients with a recent history or current signs or symptoms, as determined by the Investigator, of severe, progressive viral or bacterial infections, of clinically significant cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic insufficiency disease (excluding psoriasis) requiring systemic treatment or other major diseases, which are not well controlled and may interfere with the conduct of the trial.
9. Patients with active malignancy or history of malignancy, except for basal cell or squamous cell carcinoma and actinic keratosis. Basal cell carcinoma and small squamous cell carcinoma of the skin which have been excised according to guidelines within the last 5 years or in situ cervical carcinoma that has been fully treated and shows no evidence of recurrence are allowed.
10. Clinically significant abnormality on 12-lead electrocardiogram (ECG) at screening.
11. Positive human immunodeficiency virus (HIV), hepatitis B or hepatitis C laboratory result.
12. Previous strong sun exposure (eg, sea holiday) within the 28 days before study medication initiation.
13. Known photo allergy and/or experienced drug-induced photo toxicity.
14. Elective (planned) hospitalization or medical intervention preventing patient from following the protocol requirements.
15. Prior Treatment: Drug class >> Last dose prior to study medication initiation (washout period)

    Topical psoriasis medications (including, but not limited to corticosteroids, calcipotriene, topical vitamin D derivates, retinoids, coal tar) >> 14 days

    Topical immunosuppressive drugs (tacrolimus, pimecrolimus, or anthralin) >> 14 days (Exception: Non-medicated emollients, moisturizers and sunscreens will be allowed), Use of low potency topical steroids for critical areas such as the face, genitalia, and scalp may be allowed until 24 hours prior to randomization.

    Systemic treatment (non-biologic): Systemic immunosuppressant agents (eg: methotrexate, cyclosporine, azathioprine), Systemic fumarate, Systemic corticosteroids >> 28 days

    Phototherapy or photochemotherapy/photosensitizing drugs >> 28 days

    Systemic retinoids >> 12 weeks

    Any investigational drug >> 24 weeks (systemic); 4 weeks (topical)

    Any Anti-TNFs: Infliximab, adalimumab, golimumab, etanercept, etc. >> 12 weeks

    Other Biologics and other systemic therapies: ustekinumab, alefacept, apremilast, Efalizumab, certolizumab pegol, secukinumab, etc. >> 24 weeks

    Rituximab >> 12 months
16. Drinking or ingesting grapefruit, pomegranate, grapefruit juice or grapefruit containing products within 14 days of study medication initiation.
17. Planned use of any ultraviolet (UV) phototherapy or photochemotherapy/photosensitizing drugs during the course of the study and within 28 days following the last dose of the study medication.
18. Patients with a history of chronic alcohol or drug abuse within 6 months of study medication initiation.
19. Patients employed by MetrioPharm or a contract research organization (CRO) involved in the clinical study.
20. Vulnerable patients (eg, patients kept in detention).
21. Patients who are unable to communicate, read and understand the local language, or who display any other condition, which, in the Investigator's opinion, makes them unsuitable for clinical study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anke Gauliard, MD, Principal Investigator — Parexel
Locations (4):
- Germany (4):
  - Rothaar Studien GmbH, Berlin
  - PAREXEL International GmbH, Klinikum Westend, Berlin
  - Klinische Forschung Dresden GmbH, Dresden
  - Gemeinschaftspraxis Prof. Dr. Vanscheidt und Dr. Ukat, Freiburg im Breisgau

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MP1032: Test Product:
  100 mg MP1032 (= 2 capsules a 50 mg) are provided orally twice daily for 42 days
  MP1032: hard gelatine capsules containing 50 mg MP1032 as active ingredient
- Placebo: Placebo:
  2 capsules of Placebo are provided orally twice daily for 42 days
  Placebo: hard gelatine capsules without active ingredient
Period: Overall Study
Arm/Group | MP1032 | Placebo
Started | 23 | 23
Completed | 22 | 22
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MP1032 | Placebo | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 23 | 45
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 18 | 17 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 23 | 23 | 46
  Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Safety - Treatment Emergent Adverse Events (TEAEs) - Number of TEAEs
Description: Number of TEAEs (Treatment Emergent Adverse Events) occured was determined by treatment group.
  Furthermore, the absolute and relative frequencies for patients with a given AE, as well as the number of events of the individual AEs that have occurred throughout the study (inclusive screening), were determined within each treatment group and system organ class. Results thereto are provided in the section "Reported Adverse Events".
  AEs are collected throughout the study. Abnormal values received from Clinical Laboratory Safety Testing (hematology, biochemistry and urinalysis on Study Days 1, 15, 29, 43, 57 and 71), Vital Signs (Systolic blood pressure, diastolic blood pressure, heart rate, tympanic body temperature and respiration rate on Study Days 1, 15, 29, 43, 57 and 71), ECG (Study Days 1, 43 and 71) and Physical Examination (Study Days 1, 43 and 71) were also handled as AE.
Time Frame: Continuously from Treatment Start until the last follow-up visit on Study Day 71
Measure: Number; unit: TEAEs
Arm/Group | MP1032 | Placebo
Number analyzed (Participants) | 23 | 23
TEAEs
  All TEAEs | 27 | 32
  Serious TEAEs | 0 | 0
  Severe TEAEs | 0 | 1
  Related TEAEs | 6 | 9
  TEAEs leading to Withdrawal | 0 | 1
  TEAEs leading to Death | 0 | 0

2. Primary Outcome: Safety - Treatment Emergent Adverse Events (TEAEs) - Number of Related TEAEs by SOC
Description: Number of related TEAEs (Treatment Emergent Adverse Events) occured by SOC (System Organ class) was determined by treatment group.
  Furthermore, the absolute and relative frequencies for patients with a given AE, as well as the number of events of the individual AEs that have occurred throughout the study (inclusive screening), were determined within each treatment group and system organ class. Results thereto are provided in the section "Reported Adverse Events".
  AEs are collected throughout the study. Abnormal values received from Clinical Laboratory Safety Testing (hematology, biochemistry and urinalysis on Study Days 1, 15, 29, 43, 57 and 71), Vital Signs (Systolic blood pressure, diastolic blood pressure, heart rate, tympanic body temperature and respiration rate on Study Days 1, 15, 29, 43, 57 and 71), ECG (Study Days 1, 43 and 71) and Physical Examination (Study Days 1, 43 and 71) were also handled as AE.
Time Frame: Continuously from Treatment Start until the last follow-up visit on Study Day 71
Measure: Number; unit: TEAEs
Arm/Group | MP1032 | Placebo
Number analyzed (Participants) | 23 | 23
TEAEs
  All related TEAEs | 6 | 9
  Gastrointestinal disorders | 0 | 3
  General disorders - Administration Site Conditions | 2 | 0
  Infections and Infestations | 2 | 3
  Nervous System Disorders | 0 | 1
  Skin and Subcutaneous Tissue Disorders | 2 | 2

3. Primary Outcome: Safety - Treatment Emergent Adverse Events (TEAEs) - Number of Patients With TEAEs
Description: Number of patients with TEAEs (Treatment Emergent Adverse Events) was determined by treatment group.
  Furthermore, the absolute and relative frequencies for patients with a given AE, as well as the number of events of the individual AEs that have occurred throughout the study (inclusive screening), were determined within each treatment group and system organ class. Results thereto are provided in the section "Reported Adverse Events".
  AEs are collected throughout the study. Abnormal values received from Clinical Laboratory Safety Testing (hematology, biochemistry and urinalysis on Study Days 1, 15, 29, 43, 57 and 71), Vital Signs (Systolic blood pressure, diastolic blood pressure, heart rate, tympanic body temperature and respiration rate on Study Days 1, 15, 29, 43, 57 and 71), ECG (Study Days 1, 43 and 71) and Physical Examination (Study Days 1, 43 and 71) were also handled as AE.
Time Frame: Continuously from Treatment Start until the last follow-up visit on Study Day 71
Measure: Count of Participants; unit: Participants
Arm/Group | MP1032 | Placebo
Number analyzed (Participants) | 23 | 23
Participants
  All TEAEs | 14 | 15
  Serious TEAEs | 0 | 0
  Severe TEAEs | 0 | 1
  Related TEAEs | 5 | 5
  TEAEs leading to Withdrawal | 0 | 1
  TEAEs leading to Death | 0 | 0

4. Primary Outcome: Safety - Treatment Emergent Adverse Events (TEAEs) - Number of Patients With Related TEAEs by SOC
Description: Number of patients with related TEAEs (Treatment Emergent Adverse Events) occured by SOC (System Organ class) was determined by treatment group.
  Furthermore, the absolute and relative frequencies for patients with a given AE, as well as the number of events of the individual AEs that have occurred throughout the study (inclusive screening), were determined within each treatment group and system organ class. Results thereto are provided in the section "Reported Adverse Events".
  AEs are collected throughout the study. Abnormal values received from Clinical Laboratory Safety Testing (hematology, biochemistry and urinalysis on Study Days 1, 15, 29, 43, 57 and 71), Vital Signs (Systolic blood pressure, diastolic blood pressure, heart rate, tympanic body temperature and respiration rate on Study Days 1, 15, 29, 43, 57 and 71), ECG (Study Days 1, 43 and 71) and Physical Examination (Study Days 1, 43 and 71) were also handled as AE.
Time Frame: Continuously from Treatment Start until the last follow-up visit on Study Day 71
Measure: Count of Participants; unit: Participants
Arm/Group | MP1032 | Placebo
Number analyzed (Participants) | 23 | 23
Participants
  All related TEAEs | 5 | 5
  Gastrointestinal disorders | 0 | 2
  General disorders - Administration Site Conditions | 2 | 0
  Infections and Infestations | 2 | 3
  Nervous System Disorders | 0 | 1
  Skin and Subcutaneous Tissue Disorders | 1 | 2

5. Primary Outcome: Pharmacokinetics (PK) - Plasma Concentrations
Description: Study Day 1 - sampling 15 minutes, 30 minutes, 1 hour and 2 hours postdose Study Days 15, 29 and 43 - only one sample was taken any time postdose (time of the last dose was recorded).
  No statistical Evaluation has been performed.
Time Frame: Study Days 1, 15, 29 and 43
Population: Participants who gave plasma for PK data and finished the study. (Data from study day 43 were not calculated since less than one-third of the individual data points were quantifiable at the nominal time point.)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MP1032
Number analyzed (Participants) | 22
ng/mL
  Day 1 - 15 minutes postdose | 190.3 (153.537)
  Day 1 - 30 minutes postdose | 162.861 (64.674)
  Day 1 - 1 hour postdose | 56.875 (30.8)
  Day 1 - 2 hours postdose | 8.677 (6.629)
  Day 15 | 211.545 (151.406)
  Day 29 | 199.652 (149.857)

6. Primary Outcome: Pharmacokinetics (PK) - Maximum Observed Concentration (Cmax)
Description: Maximum observed plasma concentration (Cmax)as observed on Day 1 with sampling times of 15 minutes, 30 minutes, 1 hour, and 2 hours postdose
Time Frame: Study Day 1
Population: PK analysis set - Per Protocol Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MP1032
Number analyzed (Participants) | 22
ng/mL | 235.585 (124.726)

7. Primary Outcome: Pharmacokinetics (PK) - Time
Description: Sampling 15 minutes, 30 minutes, 1 hour, and 2 hours postdose
  t max = Time corresponding to occurence of Cmax t last = Time of last quantifiable concentration
Time Frame: Study Day 1
Population: PK analysis set - Per Protocol Set
Measure: Median (Full Range); unit: hours
Arm/Group | MP1032
Number analyzed (Participants) | 22
hours
  t max | 0.25 [0.25 to 1.02]
  t last | 1.99 [1 to 2.05]

8. Secondary Outcome: Psoriasis Area Severity Index (PASI) - Observed PASI Values
Description: Observed PASI values. PASI is a total score computed over 4 body regions with 4 assessments ranging from 0 (no symptoms) to 4 (very marked). The total score ranges from 0 to 72.
  No formal hypothesis testing, variables are summarized by descriptive statistics (n, mean, SD, ).
Time Frame: Study Day 1, 43, 57 and 71
Population: Number of patients may vary between days due to drop outs or missing data points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MP1032 | Placebo
Number analyzed (Participants) | 23 | 23
score on a scale
  Day 1 (Treatment Start) | 16.03 (7.203) | 17.25 (7.458)
  Day 43 (End of Treatment) | 14.03 (9.509) | 14.69 (8.532)
  Day 57 (Follow Up 1): number analyzed (Participants) | 22 | 23
  Day 57 (Follow Up 1) | 15.28 (10.681) | 15.97 (8.837)
  Day 71 (Follow Up 2): number analyzed (Participants) | 22 | 23
  Day 71 (Follow Up 2) | 15.21 (10.03) | 16.09 (9.363)

9. Secondary Outcome: Psoriasis Area Severity Index (PASI) - Change From Baseline
Description: Change from Baseline (PASI value Day 43 - PASI value at Day 1) / Treatment difference on Day 43
  PASI is a total score computed over 4 body regions with 4 assessments ranging from 0 (no symptoms) to 4 (very marked). The total score ranges from 0 to 72.
  Variables will be summarized by descriptive statistics (n, mean, SD), difference between groups is analyzed via non-parametric statistical testing.
Time Frame: Study Day 1 and 43
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MP1032 | Placebo
Number analyzed (Participants) | 23 | 23
score on a scale | -2.00 (3.3994) | -2.56 (5.025)
Statistical Analysis 1: Comparison: MP1032 vs Placebo; Test type: Superiority; p = 0.8785, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.64, 95% CI 2-sided [-2.09 to 3.36]

10. Secondary Outcome: Psoriasis Area Severity Index (PASI) - PASI Percentage Change - Including Subgroup Analysis AUC2h
Description: The PASI percentage change in % at Day 29 is calculated as PASI of (Day 29 - Baseline)/Baseline*100).
  The PASI percentage change in % at Day 43 is calculated as PASI of (Day 43 - Baseline)/Baseline*100).
  Baseline = Study Day 1
  PASI is a total score computed over 4 body regions with 4 assessments ranging from 0 (no symptoms) to 4 (very marked). The total score ranges from 0 to 72.
  No formal hypothesis testing, variables are summarized by descriptive statistics (n, mean, SD).
Time Frame: Study Day 1, 29 and 43
Population: Patients of verum group were grouped into the following AUC subgroups according to AUC2h values estimated using the linear-logarithmic trapezoidal method on Day 1:
  Group 1: 6 patients with the lowest AUCs; Group 2: 5 patients with the next highest AUCs; Group 3: 6 patients with the next highest AUCs; Group 4: 5 patients with the highest AUCs.
Measure: Mean (Standard Deviation); unit: Percentage - Change from Baseline Score
Groups:
- MP1032 PK Analysis Set: Test Product:
  100 mg MP1032 (= 2 capsules a 50 mg) are provided orally twice daily for 42 days
  MP1032: hard gelatine capsules containing 50 mg MP1032 as active ingredient
  Patients from the MP1032 group who provided plasma for PK purposes and completed the study.
- AUC_2h Subgroup 1: Test Product:
  100 mg MP1032 (= 2 capsules a 50 mg) are provided orally twice daily for 42 days
  MP1032: hard gelatine capsules containing 50 mg MP1032 as active ingredient
  Subgroup 1 according to AUC2h Day 1.
- AUC_2h Subgroup 2: Test Product:
  100 mg MP1032 (= 2 capsules a 50 mg) are provided orally twice daily for 42 days
  MP1032: hard gelatine capsules containing 50 mg MP1032 as active ingredient
  Subgroup 2 according to AUC2h Day 1.
- AUC_2h Subgroup 3: Test Product:
  100 mg MP1032 (= 2 capsules a 50 mg) are provided orally twice daily for 42 days
  MP1032: hard gelatine capsules containing 50 mg MP1032 as active ingredient
  Subgroup 3 according to AUC2h Day 1.
- AUC_2h Subgroup 4: Test Product:
  100 mg MP1032 (= 2 capsules a 50 mg) are provided orally twice daily for 42 days
  MP1032: hard gelatine capsules containing 50 mg MP1032 as active ingredient
  Subgroup 4 according to AUC2h Day 1.
- Placebo PK Analysis Set: Placebo:
  2 capsules of Placebo are provided orally twice daily for 42 days
  Placebo: hard gelatine capsules without active ingredient
  Patients from the placebo group who provided plasma for PK purposes and completed the study.
Arm/Group | MP1032 PK Analysis Set | AUC_2h Subgroup 1 | AUC_2h Subgroup 2 | AUC_2h Subgroup 3 | AUC_2h Subgroup 4 | Placebo PK Analysis Set
Number analyzed (Participants) | 22 | 6 | 5 | 6 | 5 | 22
Percentage - Change from Baseline Score
  Day 29 | -18.24 (24.069) | -6.61 (25.575) | -14.74 (24.96) | -35.46 (22.891) | -15.03 (16.422) | -14.57 (21.5)
  Day 43 | -17.83 (29.853) | 3.06 (23.42) | -21.82 (38.572) | -38.31 (28.353) | -14.32 (13.466) | -15.56 (27.181)

11. Secondary Outcome: Psoriasis Area Severity Index (PASI) - PASI Percentage Change - Including Subgroup Analysis AUCt
Description: as for outcome 10
Time Frame: Study Day 1, 29 and 43
Population: Patients of verum group were grouped into the following AUC subgroups according to AUCt values estimated using the linear-logarithmic trapezoidal method on Day 1:
  Group 1: 6 patients with the lowest AUCs; Group 2: 5 patients with the next highest AUCs; Group 3: 6 patients with the next highest AUCs; Group 4: 5 patients with the highest AUCs.
Measure: Mean (Standard Deviation); unit: Percentage - Change from Baseline Score
Groups:
- AUC_t Subgroup 1: Test Product:
  100 mg MP1032 (= 2 capsules a 50 mg) are provided orally twice daily for 42 days
  MP1032: hard gelatine capsules containing 50 mg MP1032 as active ingredient
  Subgroup 1 according to AUCt Day 1.
- AUC_t Subgroup 2: Test Product:
  100 mg MP1032 (= 2 capsules a 50 mg) are provided orally twice daily for 42 days
  MP1032: hard gelatine capsules containing 50 mg MP1032 as active ingredient
  Subgroup 2 according to AUCt Day 1.
- AUC_t Subgroup 3: Test Product:
  100 mg MP1032 (= 2 capsules a 50 mg) are provided orally twice daily for 42 days
  MP1032: hard gelatine capsules containing 50 mg MP1032 as active ingredient
  Subgroup 3 according to AUCt Day 1.
- AUC_t Subgroup 4: Test Product:
  100 mg MP1032 (= 2 capsules a 50 mg) are provided orally twice daily for 42 days
  MP1032: hard gelatine capsules containing 50 mg MP1032 as active ingredient
  Subgroup 4 according to AUCt Day 1.
Arm/Group | MP1032 PK Analysis Set | AUC_t Subgroup 1 | AUC_t Subgroup 2 | AUC_t Subgroup 3 | AUC_t Subgroup 4 | Placebo PK Analysis Set
Number analyzed (Participants) | 22 | 6 | 5 | 6 | 5 | 22
Percentage - Change from Baseline Score
  Day 29 | -18.24 (24.069) | -6.61 (25.575) | -27.07 (33.055) | -25.18 (19.510) | -15.03 (16.422) | -14.57 (21.5)
  Day 43 | -17.83 (29.853) | 3.06 (23.42) | -35.88 (42.928) | -26.59 (24.922) | -14.32 (13.466) | -15.56 (27.181)

12. Secondary Outcome: Psoriasis Area Severity Index (PASI) - PASI 30 and PASI 50 - Number of Patients
Description: PASI is a total score computed over 4 body regions with 4 assessments ranging from 0 (no symptoms) to 4 (very marked). The total score ranges from 0 to 72.
  PASI 30 and PASI 50 are related to the number of patients who had at least 30% (PASI 30) or 50% (PASI 50) reduction in PASI score compared to baseline (Study Day 1).
  Variables are summarized by descriptive statistics (n, mean, SD, ). Difference between groups has been analyzed via Fisher exact test.
Time Frame: Study Day 1, 29 and 43
Population: Number of patients may vary between days due to drop outs or missing data points
Measure: Number; unit: participants
Arm/Group | MP1032 | Placebo
Number analyzed (Participants) | 23 | 23
participants
  PASI 30 - Day 29: number analyzed (Participants) | 22 | 23
  PASI 30 - Day 29 | 6 | 6
  PASI 50 - Day 29: number analyzed (Participants) | 22 | 23
  PASI 50 - Day 29 | 2 | 2
  PASI 30 - Day 43 | 8 | 5
  PASI 50 - Day 43 | 3 | 4
Statistical Analysis 1: Comparison: MP1032 vs Placebo; PASI 30 - Day 29; Test type: Superiority; p = 1, Fisher Exact
Statistical Analysis 2: Comparison: MP1032 vs Placebo; PASI 50 - Day 29; Test type: Superiority; p = 1, Fisher Exact
Statistical Analysis 3: Comparison: MP1032 vs Placebo; PASI 30 - Day 43; Test type: Superiority; p = 0.5136, Fisher Exact
Statistical Analysis 4: Comparison: MP1032 vs Placebo; PASI 50 - Day 43; Test type: Superiority; p = 1, Fisher Exact

13. Secondary Outcome: Psoriasis Area Severity Index (PASI) - PASI 30 and PASI 50 - Responder Frequency
Description: PASI is a total score computed over 4 body regions with 4 assessments ranging from 0 (no symptoms) to 4 (very marked). The total score ranges from 0 to 72.
  PASI 30 and PASI 50 are related to the number of patients (responder frequency (%)) who had at least 30% (PASI 30) or 50% (PASI 50) reduction in PASI score compared to baseline (Study Day 1).
  Variables are summarized by descriptive statistics (n, mean, SD, ).
Time Frame: Study Day 1, 29 and 43
Population: Number of patients may vary between days due to drop outs or missing data points
Measure: Number; unit: percentage of participants
Arm/Group | MP1032 | Placebo
Number analyzed (Participants) | 22 | 23
percentage of participants
  PASI 30 - Day 29 | 22.27 | 26.09
  PASI 50 - Day 29 | 9.09 | 8.7
  PASI 30 - Day 43 | 34.78 | 21.74
  PASI 50 - Day 43 | 13.04 | 17.39

14. Secondary Outcome: Physician's Global Assessment (PGA) - Observed Values and Change From Baseline
Description: PGA is the physician's global assessment of the severity of psoriasis using a 7-point scale from 0 (clear) to 6 (severe).
  No formal hypothesis testing, variables will be summarized by descriptive statistics (n, mean, SD) for absolute values and changes from baseline (Study Day 1) at Study Day 43 (End of Treatment).
Time Frame: Study Day 1 and 43
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MP1032 | Placebo
Number analyzed (Participants) | 23 | 23
score on a scale
  Day 1 (Baseline) | 4.2 (0.8) | 4.4 (0.73)
  Day 43 (End of Treatment) | 3.9 (1.32) | 4.0 (1.11)
  Change from Baseline | -0.3 (0.98) | -0.4 (0.89)

15. Secondary Outcome: Dermatology Life Quality Index (DLQI) - Observed Values and Change From Baseline.
Description: DLQI is a total score ranging from 0 (life quality is not affected) to 30 (deep impact on life quality) computed from answers to 10 questions, with each answer scored from 0 (not at all) to 3 (very much).
  No formal hypothesis testing, variables will be summarized by descriptive statistics (n, mean, SD) for absolute values and changes from baseline (Study Day 1) on end of treatment (Day 43).
Time Frame: Study Day 1 and 43
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MP1032 | Placebo
Number analyzed (Participants) | 22 | 22
score on a scale
  Day 1 (Baseline) | 8.2 (3.68) | 8.6 (5.92)
  Day 43 (End of Treatment) | 7.1 (4.66) | 7.3 (5.59)
  Change from Baseline | -1 (3.91) | -1.3 (3.51)

16. Secondary Outcome: EQ-5D 5L Visual Analogue Scale (VAS)
Description: EQ-5D (VAS) is a total score which records the patients' self-rated health status with the scale numbered 0 (worst imaginable) to 100 (best imaginable)
  No formal hypothesis testing, variables will be summarized by descriptive statistics (n, mean, SD) for absolute values and changes from baseline (Study Day 1) at end of Treatment (Study Day 43).
Time Frame: Study Day 1 and 43
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MP1032 | Placebo
Number analyzed (Participants) | 23 | 23
score on a scale
  Day 1 (Baseline) | 73.7 (16.58) | 76 (11.25)
  Day 43 (End of Treatment) | 74.8 (14.62) | 76.2 (12.48)
  Change from Baseline | 1.1 (8.14) | 0.1 (10.6)

17. Secondary Outcome: Modified Nail Psoriasis Severity Index (mNAPSI) - Observed Values and Change From Baseline
Description: mNAPSI score is a total score computed from answers to 7 questions, 3 of which can be answered with a score ranging from 0 to 3, and 4 of which can be answered with a score ranging from 0 to 1. The total score ranges from 0 to 13, the higher the score the worse the outcome.
  No formal hypothesis testing, variables will be summarized by descriptive statistics (n, mean, SD) for absolute values and changes from baseline (Study Day 1) at end of Treatment (Study Day 43).
Time Frame: Study Day 1 and 43
Population: Only patients with psoriatic nail disease were evaluated
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MP1032 | Placebo
Number analyzed (Participants) | 17 | 15
score on a scale
  Day 1 (Baseline) | 3.5 (1.37) | 4.9 (1.49)
  Day 43 (End of Treatment) | 2.8 (1.64) | 4.8 (1.78)
  Change from Baseline | -0.8 (1.48) | -0.1 (0.92)

18. Primary Outcome: Pharmacokinetics (PK) - Area Under the Curve (AUC)
Description: AUC (lin-log) - Sampling 15 minutes, 30 minutes, 1 hour, and 2 hours postdose
  AUC 2h = area under the plasma concentration-time curve from time zero to 2 hours AUC t = area under the plasma concentration-time curve from time zero to the last quantifiable concentration.
Time Frame: Study Day 1
Population: PK analysis set - Per Protocol Set
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MP1032
Number analyzed (Participants) | 22
h*ng/mL
  AUC 2h | 154.161 (67.048)
  AUC t | 139.497 (63.598)

19. Primary Outcome: Pharmacokinetics (PK) - Area Under the Curve (AUC) - Subgroups
Description: as for outcome 18
Time Frame: Study Day 1
Population: PK analysis set - Per Protocol Set was divided into 4 Subgroups based on AUC levels for AUC 2h and AUC t, respectively. All patients received test product (100 mg MP1032 (= 2 capsules a 50 mg) provided orally twice daily for 42 days)
Measure: Median (Full Range); unit: h*ng/mL
Groups:
- AUC Subgroup 1: 6 patients with the lowest AUC 2h or AUC t, respectively
- AUC Subgroup 2: 5 patients with the next highest AUC 2h or AUC t, respectively
- AUC Subgroup 3: 6 patients with the next highest AUC 2h or AUC t, respectively
- AUC Subgroup 4: 5 patients with the highest AUC 2h or AUC t, respectively
Arm/Group | AUC Subgroup 1 | AUC Subgroup 2 | AUC Subgroup 3 | AUC Subgroup 4
Number analyzed (Participants) | 6 | 5 | 6 | 5
h*ng/mL
  Subgroups AUC 2h | 84.699 [63.87 to 103.92] | 114.1 [108.97 to 123.74] | 137.246 [124.9 to 166.22] | 218.482 [206.25 to 289.74]
  Subgroups AUC t | 75.934 [63.87 to 103.92] | 114.1 [108.97 to 122.12] | 134.561 [123.13 to 166.09] | 218.482 [206.83 to 289.74]

ADVERSE EVENTS:
Time Frame: AE data were collected from Enrolment to Last Visit (Study Day 71). All in all in each patient AEs were collected over a period of approximately 2-3 months.
Arm/Group | MP1032 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 14/23 | 15/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MP1032 (N=23) | Placebo (N=23)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 1 (3)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Feeling drunk (General disorders) | 1 (1) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5) | 6 (8)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes